CLINICAL TRIAL: NCT01538290
Title: Validating Non-invasive Measurements of Central Blood Pressure in Type 2 Diabetic
Brief Title: Validating Non-invasive Measurements of Central Blood Pressure in Type 2 Diabetic Patients
Acronym: IMPRESS
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: M-20110166
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Diabetes Mellitus, Type 2; Blood Pressure
Keywords: Calibration; Validation; Transfer function; SphygmoCor; Arteriograph
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators want to validate two non-invasive devices for the determination of central blood pressure, i.e. blood pressure in the aorta (artery leaving the heart).

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus, Type 2
* Age above 18 years

Exclusion Criteria:

* Atrial fibrillation or other cardiac arrhythmia
* known stenosis of aorta or arteria subclavia/brachialis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with type 2 diabetes mellitus referred to elective coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Erik Bøtker, MD,Professor, Study Director — Aarhus University Hospital, Skejby, Department of Cardiology
Locations (1):
- Aarhus University Hospital, Skejby, Department of Cardiology, Aarhus, Denmark

REFERENCES:
- [Derived] Laugesen E, Rossen NB, Peters CD, Maeng M, Ebbehoj E, Knudsen ST, Hansen KW, Botker HE, Poulsen PL. Assessment of central blood pressure in patients with type 2 diabetes: a comparison between SphygmoCor and invasively measured values. Am J Hypertens. 2014 Feb;27(2):169-76. doi: 10.1093/ajh/hpt195. Epub 2013 Dec 4. PMID 24304654
- [Derived] Rossen NB, Laugesen E, Peters CD, Ebbehoj E, Knudsen ST, Poulsen PL, Botker HE, Hansen KW. Invasive validation of arteriograph estimates of central blood pressure in patients with type 2 diabetes. Am J Hypertens. 2014 May;27(5):674-9. doi: 10.1093/ajh/hpt162. Epub 2013 Aug 31. PMID 23996499